CLINICAL TRIAL: NCT04167124
Title: Enhancing Physical Activity Levels in Youth at Risk for Cardiovascular Disease: Evaluating a Spatio-behavioral Intervention.
Brief Title: Evaluation of a Spatio-behavioral Application
Acronym: CIRCUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Melanie Henderson, Clinical assistant professor, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIRCUIT2
Record Dates: First submitted 2018-09-26; First posted 2019-11-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- multi-sensor lifestyle intervention (Experimental)
  Interventions: Behavioral: multi-sensor lifestyle intervention

INTERVENTIONS:
Behavioral: multi-sensor lifestyle intervention

SUMMARY:
The CIRCUIT program (Centre pédiatrique d'interventions en prévention et en réadaptation cardiovasculaire) of the CHU Sainte-Justine is a multidisciplinary, personalized intervention for children with cardiovascular risk. This program includes an evaluation of the physical activity pattern using wearable sensors (accelerometer, heart rate monitor and GPS), to replace the physical activity practice of the patients in their respective real life context. The accelerometer will measure physical activity and heart rate, while the GPS will serve to obtain precise information about places visited and travels in the neighborhood. The data obtained with these tools will serve to develop indicators of the "environmental diagnosis". This information will help to personalize the intervention for each patient.

ELIGIBILITY:
Inclusion Criteria:

- Children at risk of cardiovascular disease, including children with diabetes mellitus, overweight/obesity, hypertension, dyslipidemia

Exclusion Criteria:

- Patients with physical or psychological problems that impair their ability to participate in physical activity

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2010-06-28 (Actual); Primary Completion 2012-08-30 (Actual); Study Completion 2012-08-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | Baseline
  Accelerometer measured physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada